CLINICAL TRIAL: NCT00324077
Title: A Phase I Dose Escalation Study of the Combination of Dasatinib (BMS-354825) and Imatinib in Subjects With Chronic Myeloid Leukemia in Chronic Phase
Brief Title: Phase I Study of Dasatinib (BMS-354825) and Imatinib in Subjects With Chronic Myeloid Leukemia in Chronic Phase
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Insufficient Enrollment
Sponsor: Bristol-Myers Squibb (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA180-011
Record Dates: First submitted 2006-05-09; First posted 2006-05-10 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2011-04

CONDITIONS: Myeloid Leukemia, Chronic, Chronic-Phase
Keywords: Chronic phase chronic myelogenous leukemia (CML)
MeSH Terms: conditions — Leukemia, Myeloid, Chronic-Phase | interventions — Dasatinib; Imatinib Mesylate

INTERVENTIONS:
Drug: Dasatinib in combination with imatinib

SUMMARY:
The purpose of this study is to find out whether adding a new drug, dasatinib, to imatinib is safe, and whether the combination of the two drugs will help decrease the number of cells that contain the Philadelphia chromosome.

ELIGIBILITY:
Inclusion Criteria:

* males and females, 18 or older
* chronic phase Ph+ or BCR-ABL positive CML
* current complete hematologic response to imatinib
* lack of major molecular response
* on imatinib for at least one year
* on the same imatinib dose for at least 6 months
* adequate hepatic and renal function

Exclusion Criteria:

* History of accelerated or blast phase CML
* Serious uncontrolled medical disorder or active infection
* Significant cardiovascular disease or bleeding disorder
* Concurrent use of medications at risk of causing Torsades de Pointe

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-08; Primary Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose (MTD) and recommended dose of dasatinib when combined with imatinib in chronic phase CML patients.

SECONDARY OUTCOMES:
assess safety and tolerability of dasatinib and imatinib administered in combination throughout study
identify dose limiting toxicities
characterize plasma pharmacokinetics of dasatinib and imatinib in month 1
measure major molecular response rate
measure the major cytogenetic response rate
characterize mutations in the BCR-ABL gene
evaluate progressive free survival and overall survival

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Local Institution, Los Angeles, California
  - Local Institution, San Francisco, California
  - Local Institution, New York, New York